CLINICAL TRIAL: NCT04304118
Title: Rajaie Cardiomyopathy and Myocarditis Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: registry_98118
Record Dates: First submitted 2020-01-15; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Clinical Characteristics; Natural History; Long-term Outcomes; Current Therapeutic Approaches

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of patients with cardiomyopathies who referred to Rajaei Cardiovascular medical and research center is remarkable, and also the mission of this center is to achieve center of excellence in the field of cardiomyopathy. Rajaie Cardiomyopathy and myocarditis Registry study is an observational registry of consecutive patients with four cardiomyopathy subtypes: hypertrophic cardiomyopathy (HCM), dilated cardiomyopathy (DCM), arrhythmogenic right ventricular cardiomyopathy (ARVC), and restrictive cardiomyopathy (RCM) as well as myocarditis designed to determine clinical characteristics, natural history, current therapeutic approaches, response to treatment and long-term outcomes of patients with cardiomyopathy and myocarditis and to address limitations in extant evidence to improve prognostication in cardiomyopathies and myocarditis. Prediction of mortality and response to different treatments in these patients using artificial intelligence is another aim of this registry

ELIGIBILITY:
Inclusion Criteria:

1. age greater than one year
2. documented cardiomyopathy/ myocarditis fulfilling standard diagnostic criteria
3. able to give informed consent or in the case of child consent from a parent

Exclusion Criteria:

Patients who have not consent to participate in the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with documented cardiomyopathy/ myocarditis fulfilling standard diagnostic criteria based on the ESC guideline for cardiomyopathy/ myocarditis
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-11-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Admissions to hospital | 1 year
  Number of hospitalizations for cardiovascular reasons
Development of chronic heart failure | 1 year
  significant decrease in left ventricular ejection fraction
Prevalence of Stroke/Transient ischemic attack | 1 year
  At least 80% CT/MRI verification of the diagnosis of ischemic stroke/Transient ischemic attack, within the first week of stroke onset
Incidence of sudden death | 1 year
  unexpected death from a cardiovascular cause in a person with or without preexisting heart disease
Incidence of heart trasplantation | 1 year
  Cardiac transplantation in patients with end-stage HF who remain symptomatic despite optimal medical therapy

SECONDARY OUTCOMES:
response to current therapeutic approaches | 1 year
  Implantable cardioverter defibrillator implantation, Cardiac resynchronisation therapy, septal myectomy, ablation, cardiac transplantation and medications

CONTACTS AND LOCATIONS:
Locations (1):
- Behshid Ghadrdoost, Tehran, Iran